CLINICAL TRIAL: NCT00210639
Title: A Multicenter, Long-Term, Active-Surveillance Study of Musculoskeletal Disorders That Occur After Initiating a Course of Levofloxacin (RWJ-25213-097) or Non-Fluoroquinolone Therapy for Acute Infectious Diseases in Children Who Were Enrolled in Phase 3 Clinical Trials Involving Levofloxacin Therapy
Brief Title: A Study of Incidence of Musculoskeletal Disorders in Children Who Have Received Levofloxacin or a Standard Non-Fluoroquinolone Therapy for Acute Bacterial Infection
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004171; LOFBO-LTSS-001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); PRI/LOF-INT-4 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Musculoskeletal Diseases
Keywords: Musculoskeletal Diseases; Musculoskeletal Disorders; Childhood Disease; Bone Diseases; Joint Diseases; Levofloxacin; Quinolones; Bacterial infections
MeSH Terms: conditions — Musculoskeletal Diseases; Bone Diseases; Joint Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Levofloxacin-treated cohort: Participants receiveing levofloxacin in previous levofloxacin studies will be observed.
  Interventions: Drug: No intervention
- Comparator-treated cohort: Participants receiveing comparator in previous levofloxacin studies will be observed.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Participants rceiving dosing regimen from the respective Phase 3 levofloxacin clinical studies will be observed in this study.

SUMMARY:
The purpose of this study is to assess the long-term safety of levofloxacin administered to children as therapy for acute bacterial infection.

DETAILED DESCRIPTION:
This is a prospective (look forward using periodic observations collected predominantly following participant enrollment), long-term, comparative, multicenter, observational study (study in which the investigators/physicians observe the participants and measure their outcomes) to monitor long-term the incidence of musculoskeletal (MS) disorders in children who have received levofloxacin or a standard therapy for acute bacterial infection. Approximately 2500 participants who were enrolled in prior Phase 3 clinical studies of the use of levofloxacin for the treatment of acute infectious disease will be observed in this study. The study consists of 3 phases: a screening phase; a surveillance phase; and a musculoskeletal disorder follow-up phase. Safety evaluations will include assessment of an overall incidence of musculoskeletal disorders that occur during the first 60 days after the first dose of anti-microbial therapy. The specific musculoskeletal disorders to be reported are: tendinopathy (inflammation or rupture of a tendon); arthritis (inflammation of a joint as shown by redness or swelling); arthralgia (pain in a joint); gait abnormality (limping or refusal to walk). Other assessments of safety will include interviews using standardized questionnaires to assess the occurrence of musculoskeletal adverse events, physical examinations, and measurement of participants height over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Must have taken at least 1 dose of levofloxacin or standard non-fluoroquinolone therapy as part of a Phase 3 levofloxacin clinical study (LOFBIV-PCAP-003, LOFBO-OTMD-001, LOFBO-OTMD-002) to treat an acute bacterial infection
* Parent or legal guardian read and signed the informed consent form

Exclusion Criteria:

* Participants who do not meet the criteria for enrollment in a prior Phase 3 clinical study of levofloxacin or did not take at least one dose of levofloxacin or standard non-fluoroquinolone therapy in 1 of 3 prior Phase 3 levofloxacin clinical studies (LOFBIV-PCAP-003, LOFBO-OTMD-001, or LOFBO-OTMD-002)

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who have received levofloxacin or a standard non-fluoroquinone therapy for acute bacterial infection in one of the Phase 3 interventional studies will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 2233 (Actual)
Dates: Start 2002-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L .C.Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (62):
- United States (47):
  - Hoover, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Madera, California
  - Oakland, California
  - Orange, California
  - Paramount, California
  - San Luis Obispo, California
  - West Covina, California
  - Centennial, Colorado
  - Denver, Colorado
  - Chiefland, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Blue Ridge, Georgia
  - Marietta, Georgia
  - ‘Aiea, Hawaii
  - Boise, Idaho
  - Nampa, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Bardstown, Kentucky
  - Louisville, Kentucky
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Slidell, Louisiana
  - Detroit, Michigan
  - Royal Oak, Michigan
  - Stevensville, Michigan
  - Omaha, Nebraska
  - Johnson City, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Corpus Christi, Texas
  - Houston, Texas
  - Seguin, Texas
  - Burke, Virginia
  - Vienna, Virginia
- Argentina (3):
  - Buenos Aires
  - Loma Hermosa
  - San Isidro
- Brazil (3):
  - Curitiba
  - Porto Alegre
  - São Paulo
- Santiago, Chile
- Costa Rica (2):
  - Costa Rica
  - San José
- Beersheba, Israel
- Mexico (4):
  - Guadalajara
  - Puebla City
  - Toluca
  - Zapopan
- Zona, Panama

REFERENCES:
- [Result] Noel GJ, Bradley JS, Kauffman RE, Duffy CM, Gerbino PG, Arguedas A, Bagchi P, Balis DA, Blumer JL. Comparative safety profile of levofloxacin in 2523 children with a focus on four specific musculoskeletal disorders. Pediatr Infect Dis J. 2007 Oct;26(10):879-91. doi: 10.1097/INF.0b013e3180cbd382. PMID 17901792
- [Derived] Bradley JS, Kauffman RE, Balis DA, Duffy CM, Gerbino PG, Maldonado SD, Noel GJ. Assessment of musculoskeletal toxicity 5 years after therapy with levofloxacin. Pediatrics. 2014 Jul;134(1):e146-53. doi: 10.1542/peds.2013-3636. Epub 2014 Jun 2. PMID 24918220
- See also: A long-term study of the incidence of musculoskeletal disorders in children who have received levofloxacin or a standard non-fluoroquinolone therapy for acute bacterial infection — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=57&filename=CR004171_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, a total of 2233 participants were enrolled; 1620 participants from 2 otitis media studies (LOFBO-OTMD-001, LOFBO-OTMD-002) and 613 from a community acquired pneumonia study (LOFBIV-PCAP-003).
Pre-assignment Details: Only 207 participants out of 2233 participants were required for yearly follow-up during the Musculoskeletal Disorder (MSD) follow-up phase.
Groups:
- Levofloxacin: Participants who received levofloxacin in the previous studies.
- Comparator: Participants who received comparator in the previous studies.
Period: Overall Study
Arm/Group | Levofloxacin | Comparator
Started | 124 | 83
Completed | 61 | 41
Not Completed | 63 | 42
Not completed — Lost to Follow-up | 37 | 29
Not completed — Withdrawal by Subject | 8 | 1
Not completed — Other | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin | Comparator | Total
Number analyzed (Participants) | 124 | 83 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.9 (2.52) | 3.5 (2.46) | 3.7 (2.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 76 | 43 | 119
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 16 | 11 | 27
  BRAZIL | 8 | 4 | 12
  CHILE | 10 | 12 | 22
  COSTA RICA | 27 | 15 | 42
  ISRAEL | 2 | 0 | 2
  MEXICO | 0 | 1 | 1
  PANAMA | 0 | 1 | 1
  UNITED STATES | 61 | 39 | 100
AgeCategorical [Number; unit: participants]
  <2 YEARS | 16 | 14 | 30
  2-<6 YEARS | 95 | 62 | 157
  6-<12 YEARS | 9 | 5 | 14
  12-<17 YEARS | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Musculoskeletal Adverse Events During the Musculoskeletal Disorder Follow-up Phase
Description: The criteria used to assess Musculoskeletal Adverse Event is based on system organ class "Musculoskeletal and connective tissue disorders" of MedDRA 13.0.
Time Frame: Musculoskeletal Disorder (MSD) Follow-Up phase (ie, up to 5 years after their first dose of antimicrobial therapy, yearly visits for 4 additional years)
Population: Participants (207) who were followed up during the MSD Follow-Up Phase.
Measure: Number; unit: Participants
Arm/Group | Levofloxacin | Comparator
Number analyzed (Participants) | 124 | 83
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Levofloxacin | Comparator
Serious Adverse Events (participants affected / at risk) | 2/124 | 3/83
Other Adverse Events (participants affected / at risk) | 3/124 | 6/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=124) | Comparator (N=83)
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Otitis Media Chronic (Infections and infestations) | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levofloxacin (N=124) | Comparator (N=83)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypermobility Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral Pain Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 2
Spastic Paralysis (Nervous system disorders) | 0 | 1
Otoplasty (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
This was an observational safety study with no efficacy endpoints. Adverse event data is entered into the appropriate section within this submission.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days